CLINICAL TRIAL: NCT06478927
Title: A Single-Arm, Prospective, Open Clinical Study of Palbociclib for Backline Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Backline Treatment of Advanced Hepatocellular Carcinoma With Palbociclib
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-HCC-Palbociclib-001
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — palbociclib

STUDY DESIGN:
Intervention Model Description: Palbociclib Capsules
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palbociclib Group (Experimental): Palbociclib capsules, oral, qd
  Interventions: Drug: Palbociclib capsules

INTERVENTIONS:
Drug: Palbociclib capsules — Palbociclib capsules, oral, 125 mg/dose, qd, take 3 weeks and then stop for 1 week, 28d for one treatment cycle until disease progression or intolerable toxicity.
  Other Names: Palbociclib

SUMMARY:
Currently, it has been demonstrated that CDK4 is highly expressed in hepatocellular carcinoma patients and is significantly associated with poor prognosis in hepatocellular carcinoma patients. Palbociclib is the world's first marketed inhibitor of the cell cycle protein-dependent kinase CDK4/6, which is capable of blocking cell cycle progression and inhibiting tumor cell proliferation. However, current evidence for the use of CDK4/6 inhibitors in patients with advanced hepatocellular carcinoma cells remains lacking. This study used palbociclib backline treatment for patients with advanced hepatocellular carcinoma, aiming to further validate the potential role of CDK4/6 inhibitors in the treatment of patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
This study was a single arm, prospective, open clinical study. Twenty-two patients with advanced hepatocellular carcinoma were enrolled in this study and were simultaneously treated and observed with palbociclib. The efficacy and safety of palbociclib in patients with advanced hepatocellular carcinoma were evaluated by PFS, ORR, DCR, OS, and AE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years and ≤75 years;
2. ECOG score 0~2;
3. Patients with histologically or cytologically confirmed unresectable advanced hepatocellular carcinoma;
4. Patients who have failed or are intolerant of at least second-line treatment;
5. Expected survival ≥ 3 months;
6. An evaluable lesion within 21 days prior to enrollment according to RECIST 1.1 criteria;
7. Barcelona Clinical Liver Cancer Staging (BCLC staging) stage B or C and not suitable for surgical or local treatment, or progression after surgery or local treatment;
8. Child-Pugh Liver Function Class: Grade A or B (≤7 points);
9. HBV DNA quantification must be <500IU/ml or 2500 copies/ml and receive at least 2 weeks of anti-HBV treatment before study entry; HCVRNA quantification-positive patients must have completed antiviral treatment at least 1 month before study entry;
10. CNS metastases without clinical symptoms or with clinical symptoms controlled and stabilized for ≥4 weeks after treatment：

(1) Routine blood tests should meet the following criteria: ANC ≥1.0×109/L; PLT ≥50×109/L; Hb ≥80 g/L; (2) Biochemical tests must meet the following criteria: TBIL ≤ 3 times the upper limit of normal (ULN); ALT and AST ≤ 5 times the upper limit of normal (ULN); serum creatinine ≤ 1.5 × ULN or creatinine clearance rate > 50 ml/min (Cockcroft-Gault formula); (3) Coagulation examination criteria to be met: prothrombin time (PT) ≤ 1.5 x ULN, activated partial thromboplastin kinase time (aPTT) ≤ 1.5 x ULN; (4) Cardiac ultrasound and echocardiography: left ventricular ejection fraction (LVEF ≥ 55%), ECG QTc < 450ms (men), QTc < 470ms (women); 13. Patients who agree to abstain from sex or use an effective method of contraception for the duration of treatment and for at least 7 months after the last dose of study treatment; 14. Signed informed consent.

Exclusion Criteria:

1. Prior treatment with any CDK4/6 inhibitor drug;
2. Patient has received antitumor therapy in another clinical trial within 4 weeks prior to enrollment;
3. Patient has undergone a major surgical operation within 4 weeks prior to enrollment or the patient has not fully recovered from such surgical operation;
4. Severe cardiac disease or discomfort;
5. Hepatitis B combined with Hepatitis C or Hepatitis D infection;
6. Patient is allergic to the components of the drug perphenazine or its excipients;
7. Other malignant tumors within 5 years (except cured basal cell carcinoma of the skin, carcinoma in situ of the prostate and carcinoma in situ of the cervix);
8. Those with multiple factors affecting the oral administration of drugs (e.g. inability to swallow, post gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.);
9. Pregnant or breastfeeding female patients, female patients of childbearing potential with a positive baseline pregnancy test, or patients of childbearing potential who are unwilling to use effective contraception throughout the trial period and for 7 months after the final study dose;
10. Severe concomitant disease or other co-morbidities that would interfere with planned therapy, or any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to approximately 2 years.
  PFS is defned as the time from randomization untlthe date of first occurence of investigator assessed radiolbgical disease progression or death due to any cause,whichever came first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to approximately 2 years.
  ORR is defied as the percentage of subject with complete response (CR) or partial response (PR) by investigator assessment per REclsT criteria, version 1.1.
Disease control rate (DCR) | up to approximately 2 years.
  DCR was defined as the percentage of patients who have achieved complete response (CR), partial response (PR) and stable disease (SD).
Overall survival (OS) | up to approximately 2 years.
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Adverse Events (AE) | up to approximately 2 years.
  AE assessed by NCI-CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zhuang, M.D., Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No